CLINICAL TRIAL: NCT05461352
Title: A Multi-center, Open-label Long-Term Study of TS-142 in Patients with Insomnia Disorder
Brief Title: Long-Term Study of TS-142 in Patients with Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TS142-302
Record Dates: First submitted 2022-07-07; First posted 2022-07-18 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-03

CONDITIONS: Patients with Insomnia
MeSH Terms: interventions — TS-142

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5 mg (Experimental): Period in which participants received repeated doses of 5 mg TS-142 prior to bedtime
  Interventions: Drug: TS-142 5 mg
- 10 mg (Experimental): Period in which participants received repeated doses of 10 mg TS-142 prior to bedtime
  Interventions: Drug: TS-142 10 mg

INTERVENTIONS:
Drug: TS-142 5 mg — Participants received repeated doses of 5 mg of TS-142 (oral tablet)
  Arms: 5 mg
Drug: TS-142 10 mg — Participants received repeated doses of 10 mg of TS-142 (oral tablet)
  Arms: 10 mg

SUMMARY:
This is a randomized, open-label, multi-center long-term study in patients with insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese male and female who are aged 18 years or older at the time of informed consent
2. Outpatients
3. Patients falling under the category of insomnia disorder according to the diagnostic criteria in the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5)

Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

1. Patients falling under the category of any disorders other than insomnia disorder among sleep-wake disorders according to the diagnostic criteria in DSM-5
2. Patients with psychiatric diseases other than depression and anxiety
3. Patients with symptoms such as pain, pruritus, frequent urination and asthma that seriously prevent their sleep

Other protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | From start of investigational drug administration to final test and observation; up to approximately 1 year
  To evaluate the Long-term safety of TS-142 in patients with insomnia

SECONDARY OUTCOMES:
Mean change from baseline of subjective sleep latency (sSL) | From baseline up to Week 52
  sSL defined as the duration of time that it took to fall asleep as recorded in a sleep diary.
Mean change from baseline of subjective sleep efficacy (sSE) | From baseline up to Week 52
  sSE is defined as the percentage of total sleep time (TST) in total amount of time from bedtime to wake-up time in a sleep diary.
Mean change from baseline of subjective total sleep time (sTST) | From baseline up to Week 52
  sTST defined as the total amount of time spent asleep before wake-up time as recorded in a sleep diary.
Mean change from baseline of subjective wake time after sleep onset (sWASO) | From baseline up to Week 52
  sWASO is defined as the total amount of time spent awake after falling asleep and before wake-up time as recorded in a sleep diary.
Mean change from baseline of subjective number of awakenings (sNAW) | From baseline up to Week 52
  sNAW is defined as the total number of awaking after falling asleep and before getting out of bed as recored in a sleep diary

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No